CLINICAL TRIAL: NCT07003308
Title: Comparative Study of the Efficacy of Anterior Versus Posterior White Line Advancement Technique in the Correction of Primary Aponeurotic Ptosis
Brief Title: Anterior Versus Posterior White Line Advancement Technique in the Correction of Aponeurotic Ptosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Viviana Patricia Lezcano Carduz, Principal Investigator., Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC054-25_HRJC
Record Dates: First submitted 2025-05-06; First posted 2025-06-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-05

CONDITIONS: Ptosis, Eyelid
Keywords: eyelid; levator palpebrae; oculoplastic surgery; ophthalmology; blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Approach Group (Experimental): Participants will undergo upper eyelid ptosis correction using the anterior approach, involving a skin incision through the upper eyelid crease to access the levator aponeurosis
  Interventions: Procedure: Anterior White Line Advancement Surgery
- Posterior Approach Group (Active Comparator): Participants will undergo upper eyelid ptosis correction using the posterior approach, which avoids skin incision and accesses the levator aponeurosis via the conjunctiva.
  Interventions: Procedure: Posterior White Line Advancement Surgery

INTERVENTIONS:
Procedure: Anterior White Line Advancement Surgery — This technique involves a skin incision at the eyelid crease, dissection through the orbicularis muscle to expose the tarsus, and proximal dissection in the pre-Müller-conjunctival plane to visualize the white line. A double-armed 5-0 absorbable suture is used to advance the white line to the anterior tarsal surface. Eyelid height and contour are assessed before final fixation. Skin closure is completed with a non-absorbable suture.
  Arms: Anterior Approach Group
Procedure: Posterior White Line Advancement Surgery — This conjunctival technique uses a traction suture and eyelid eversion to access the posterior surface of the eyelid. A conjunctival incision is made above the superior tarsal border, followed by dissection to expose the white line. A double-armed 5-0 absorbable suture is passed through the anterior tarsus and the white line, and tied after confirming adequate eyelid position. The conjunctiva is not sutured.
  Arms: Posterior Approach Group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two surgical techniques-anterior and posterior white line advancement-for the correction of primary aponeurotic ptosis in adult patients. The main questions it aims to answer are:

Does the anterior approach lead to a greater improvement in Marginal Reflex Distance 1 (MRD1) at 6 months compared to the posterior approach?

Are there differences in eyelid symmetry, contour, visual function, and patient satisfaction between the two techniques?

Researchers will compare the anterior approach group to the posterior approach group to see if one offers better functional and aesthetic outcomes, fewer complications, or higher patient satisfaction.

Participants will:

Be randomly assigned to receive either anterior or posterior white line advancement surgery.

Undergo preoperative and postoperative evaluations at 7 days, 2 months, and 6 months, including:

Measurements of eyelid position (MRD1), contour, and symmetry

Vision and tear film tests (e.g., refraction, TBUT, Schirmer's test)

Surveys on dry eye symptoms (OSDI), scar quality (POSAS 2.0), satisfaction, and psychosocial function

Monitoring of surgical time and complications

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical trial designed to compare the efficacy, functional outcomes, aesthetic results, and patient-reported satisfaction associated with two surgical techniques for correcting primary aponeurotic ptosis: anterior white line advancement and posterior white line advancement.

Participants will be randomized 1:1 into two parallel groups. In the anterior approach, access to the levator aponeurosis is achieved via a skin crease incision, and advancement is performed using sutures placed on the white line to reattach it to the anterior surface of the tarsus. In the posterior approach, access is gained through a conjunctival incision above the superior tarsal border, followed by dissection to expose the white line and suture advancement to the anterior tarsus, without a skin incision.

Functional eyelid position will be assessed through MRD1 measurements, symmetry evaluation, and contour analysis. Contour will be quantified objectively using ImageJ software with Bézier curve fitting, and subjectively through independent masked evaluations based on pre-defined criteria.

Patient-reported outcomes will be assessed using the validated FACE-Q Aesthetics questionnaire, including scales for appearance satisfaction, psychosocial function, early recovery, and satisfaction with the surgical outcome and decision. Tear film stability and ocular surface parameters will be assessed using TBUT, Schirmer test (without anesthesia), and the Ocular Surface Disease Index (OSDI).

Standardized digital photographs will be taken at each follow-up visit to ensure consistent evaluation of eyelid contour and aesthetic results. All images and clinical data will be securely stored with restricted access for authorized investigators only.

Follow-up visits are scheduled for Day 7, Month 2, and Month 6 postoperatively. No masking will be applied due to the nature of the surgical techniques; however, outcome assessors for eyelid contour and patient-reported measures will remain blinded to group assignment.

This study aims to generate high-quality comparative data to guide clinical decision-making in the surgical management of aponeurotic ptosis, with an emphasis on both anatomical and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Diagnosis of primary aponeurotic upper eyelid ptosis.
* Levator muscle function of 12 mm or greater.
* Provision of written informed consent after receiving adequate information about the study.

Exclusion Criteria:

* Diagnosis of non-aponeurotic eyelid ptosis.
* Poor levator muscle function.
* History of recurrent eyelid ptosis or previous eyelid ptosis surgery.
* Medical or surgical history that, in the investigator's judgment, may interfere with participation.
* Individuals with childbearing potential who are not using highly effective contraception methods.
* Refusal to participate in the study or to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Marginal Reflex Distance 1 (MRD1) at 6 Months | Baseline (Day 0) and Month 6 (±2 weeks) after surgery
  MRD1 will be measured preoperatively and at 6 months postoperatively to assess the difference in eyelid position between the anterior and posterior approach groups.

SECONDARY OUTCOMES:
Change in MRD1 at 2 Months | Baseline (Day 0) and Month 2 (±1 week) after surgery
  Measured preoperatively and at 2 months postoperatively to compare eyelid position between groups.
Postoperative Interpalpebral Symmetry at 2 and 6 Months | Month 2 (±1 week) and Month 6 (±2 weeks) after surgery
  Symmetry between eyelids will be evaluated to assess aesthetic outcomes.
Eyelid Contour Evaluation at 2 and 6 Months | Month 2 (±1 week) and Month 6 (±2 weeks) after surgery
  Eyelid contour will be assessed using standardized frontal photographs in primary gaze.
  Objective analysis will be performed with ImageJ software using the Bézier plugin to calculate the percentage of overlap with an ideal curve (Excellent: >90%, Good: 85-90%, Poor: <85%).
  Subjective assessment will be conducted by three masked investigators based on symmetry, curvature, and slope criteria, rated as Excellent (3/3), Good (2/3), or Poor (0-1/3).
Change in Refractive Error at 2 and 6 Months | Baseline (Day 0), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Comparison of pre- and postoperative refractive measurements.
Change in Corneal Topographic Parameters at 2 and 6 Months | Baseline (Day 0), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Assessed using corneal topography to evaluate changes related to surgery.
Change in Tear Break-Up Time (TBUT) at 2 and 6 Months | Baseline (Day 0), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Measured to assess the impact on tear film stability. TBUT will be measured by instilling fluorescein dye and recording the time (in seconds) from the last blink to the first appearance of a dry spot on the cornea. Each eye will be assessed three times, and the mean value will be used. Lower values indicate greater tear film instability. A TBUT <10 seconds is considered abnormal.
Change in Schirmer Test (without anesthesia) at 2 and 6 Months | Baseline (Day 0), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Evaluates tear production before and after surgery. The Schirmer I test (without anesthesia) measures basal and reflex tear production. Standardized strips will be placed in the lower fornix for 5 minutes. The length of wetting (in mm) will be recorded. Values <10 mm indicate decreased tear production.
Change in Ocular Surface Disease Index (OSDI) Scores at 7 Days, 2 and 6 Months | Baseline (Day 0), Day 7 (±1 day), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Patient-reported outcomes on dry eye symptoms. The OSDI questionnaire includes 12 items assessing symptoms, visual function, and environmental triggers. Raw scores are converted to a 0-100 scale using the formula: (sum of scores × 25) ÷ number of questions answered. Higher scores indicate greater symptom severity. Classification: 0-12 (normal), 13-22 (mild), 23-32 (moderate), ≥33 (severe).
Change in Aesthetic Satisfaction Scores at 2 Months | Baseline (Day 0) and Month 2 (±1 week) after surgery
  Assessed with the FACE-Q Aesthetics "Satisfaction with Eyes" scale. Raw scores are summed and converted to a 0-100 scale using the official Conversion Table. If ≥50% of items are answered, missing values are imputed using the within-person mean. Higher scores indicate greater satisfaction.
Change in Psychosocial Function Scores at 2 Months | Baseline (Day 0) and Month 2 (±1 week) after surgery
  Patient-reported impact of surgery on self-image and social interaction. Measured using FACE-Q Aesthetics scales: Psychological Function, Social Function, and Appearance-Related Distress. Raw scores are summed and converted (0-100). Imputation is applied when ≥50% of items are answered. Higher scores reflect better outcomes, except for Distress, where higher scores indicate worse distress.
Assessment of Early Symptom Recovery at 7 Days | Day 7 (±1 day) after surgery
  Evaluates discomfort, swelling, and return to normal activities. Assessed with FACE-Q Aesthetics scales for "Recovery Early Symptoms" and "Eyelids-upper." Scoring follows standard FACE-Q procedure with 0-100 conversion. Missing values are imputed if ≥50% of items are answered. Higher scores reflect better recovery and appraisal.
Satisfaction with Surgical Outcome and Decision at 2 Months | Month 2 (±1 week) after surgery
  Includes willingness to undergo the procedure again. Evaluated using FACE-Q Aesthetics scales: "Satisfaction with Outcome" and "Satisfaction with Decision." Scores range from 0 (worst) to 100 (best). Missing data is managed per FACE-Q guidelines: impute mean values if ≥50% of items are completed.
Incidence of Surgical Complications Using Clavien-Dindo Classification | Day of surgery (Day 0), Day 7 (±1 day), Month 2 (±1 week), and Month 6 (±2 weeks) after surgery
  Surgical complications recorded intraoperatively, and at 7 days, 2 and 6 months.
Surgical Time Comparison | Day of surgery (Day 0); from operating room entry to exit (recorded in minutes)
  Total duration of the surgical procedure, defined as the time elapsed from the patient's entry into the operating room until their exit after completion of surgery, will be recorded and compared between each surgery group.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Patricia Lezcano Carduz, MD, Principal Investigator — Rey Juan Carlos Hospital
Locations (1):
- Rey Juan Carlos Hospital, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns related to patient confidentiality and data protection regulations

REFERENCES:
- [Background] Shen Y, Yu W, Ding F, Lu L, Liu F, Sun D, Luo X, Jin R, Yang J. Aesthetic Correction of Mild-to-Moderate Blepharoptosis Among Asians: The Bridge Technique. Ophthalmol Ther. 2022 Feb;11(1):151-160. doi: 10.1007/s40123-021-00417-3. Epub 2021 Nov 6. PMID 34741757
- [Background] Ozturk Karabulut G, Fazil K. Corneal Topographical Changes After Muller's Muscle-conjunctival Resection Surgery. Ophthalmic Plast Reconstr Surg. 2019 Mar/Apr;35(2):177-181. doi: 10.1097/IOP.0000000000001203. PMID 30130332
- [Background] Inal Ozen M, Demirok G, Yalniz Akkaya Z, Akbas Kocaoglu F, Katircioglu Y, Celik T, Ornek F, Acar DD. Effect of upper eyelid blepharoplasty surgery on cornea biomechanics and ocular surface. Int Ophthalmol. 2024 Sep 22;44(1):386. doi: 10.1007/s10792-024-03313-4. PMID 39306627
- [Background] Aksu Ceylan N, Yeniad B. Effects of Upper Eyelid Surgery on the Ocular Surface and Corneal Topography. Turk J Ophthalmol. 2022 Feb 23;52(1):50-56. doi: 10.4274/tjo.galenos.2021.63255. PMID 35196840
- [Background] Bilici S, Harbigil-Sever T, Ugurbas SH. Digital analysis of unilateral ptosis repair: external levator advancement vs. Muller's muscle conjunctival resection. Arq Bras Oftalmol. 2024 Mar 22;87(3):e20230028. doi: 10.5935/0004-2749.2023-0028. eCollection 2024. PMID 38537045
- [Background] Schulz CB, Nicholson R, Penwarden A, Parkin B. Anterior approach white line advancement: technique and long-term outcomes in the correction of blepharoptosis. Eye (Lond). 2017 Dec;31(12):1716-1723. doi: 10.1038/eye.2017.138. Epub 2017 Aug 11. PMID 28799556
- [Background] Patel V, Salam A, Malhotra R. Posterior approach white line advancement ptosis repair: the evolving posterior approach to ptosis surgery. Br J Ophthalmol. 2010 Nov;94(11):1513-8. doi: 10.1136/bjo.2009.172353. Epub 2010 Sep 10. PMID 20833687
- [Background] Sagili S. Anterior Approach White-Line Advancement: A Hybrid Technique for Ptosis Correction. Ophthalmic Plast Reconstr Surg. 2015 Nov-Dec;31(6):478-81. doi: 10.1097/IOP.0000000000000543. PMID 26325380
- [Background] Mangan MS, Cakir A, Imamoglu S. Cumulative Sum Analysis of the Learning Curve of Ptosis Surgery: External Levator Advancement versus Muller Muscle-conjunctival Resection. Korean J Ophthalmol. 2021 Oct;35(5):383-390. doi: 10.3341/kjo.2021.0058. Epub 2021 Aug 3. PMID 34344132
- [Background] Arslan N, Bahar A, Acar M, Kosker M, Kabatas N, Gurdal C. The results of Muller Muscle Conjunctival Resection versus Levator Advancement for mild to moderate ptosis. Rom J Ophthalmol. 2023 Apr-Jun;67(2):128-133. doi: 10.22336/rjo.2023.23. PMID 37522026
- [Background] Antus Z, Salam A, Horvath E, Malhotra R. Outcomes for severe aponeurotic ptosis using posterior approach white-line advancement ptosis surgery. Eye (Lond). 2018 Jan;32(1):81-86. doi: 10.1038/eye.2017.128. Epub 2017 Aug 4. PMID 28776587
- [Background] Habroosh FA, Eatamadi H. Conjunctival Sparing Ptosis Correction by White-Line Advancement Technique. J Ophthalmol. 2020 Jul 15;2020:9021848. doi: 10.1155/2020/9021848. eCollection 2020. PMID 32733700
- [Background] Kim KK, Granick MS, Baum GA, Beninger F, Cahill KV, Donnelly KC, Kaidi AA, Kang AS, Loeding L, Loyo M, Patel PA, Roostaeian J, Taghva GH, Varkarakis GM. American Society of Plastic Surgeons Evidence-Based Clinical Practice Guideline: Eyelid Surgery for Upper Visual Field Improvement. Plast Reconstr Surg. 2022 Aug 1;150(2):419e-434e. doi: 10.1097/PRS.0000000000009329. Epub 2022 Jul 27. PMID 35895522
- [Background] Karam M, Alsaif A, Abul A, Alkhabbaz A, Alotaibi A, Shareef E, Behbehani R. Muller's muscle conjunctival resection versus external levator advancement for ptosis repair: systematic review and meta-analysis. Int Ophthalmol. 2023 Jul;43(7):2563-2573. doi: 10.1007/s10792-023-02633-1. Epub 2023 Jan 24. PMID 36692699
- [Background] Bacharach J, Lee WW, Harrison AR, Freddo TF. A review of acquired blepharoptosis: prevalence, diagnosis, and current treatment options. Eye (Lond). 2021 Sep;35(9):2468-2481. doi: 10.1038/s41433-021-01547-5. Epub 2021 Apr 29. PMID 33927356
- [Background] Kakizaki H, Zako M, Nakano T, Asamoto K, Miyaishi O, Iwaki M. The levator aponeurosis consists of two layers that include smooth muscle. Ophthalmic Plast Reconstr Surg. 2005 Sep;21(5):379-82. PMID 16234705